CLINICAL TRIAL: NCT06560892
Title: Comparison Between Mean Duration of Post-operative Analgesia of Intraperitoneal Bupivacaine Alone or With Dexmedetomidine Following Laparoscopic Cholecystectomy
Brief Title: Comparison of Intraperitoneal Bupivacaine Alone or With Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Collaborators: Bahawal Victoria Hospital (Unknown)
Responsible Party: Principal Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DRQAZIANEESBVH
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: LAPAROSCOPIC CHOLECYSTECTOMY
MeSH Terms: interventions — Bupivacaine; Anesthetics, Local; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine group (Experimental): Patients received intraperitoneal bupivacaine 50 ml 0.25% + 5 ml normal saline
  Interventions: Drug: Bupivacaine injection
- Bupivacaine + Dexmedetomidine group (Experimental): Patients were given intraperitoneal bupivacaine 50 ml 0.25% + dexmedetomidine 1 μg/kg with normal saline 5 ml
  Interventions: Drug: Bupivacaine injection; Drug: Dexmedetomidine injection

INTERVENTIONS:
Drug: Bupivacaine injection — patients received intraperitoneal bupivacaine 50 ml 0.25% + 5 ml normal saline.
  Other Names: Local anesthetic
Drug: Dexmedetomidine injection — Patients were given intraperitoneal bupivacaine 50 ml 0.25% + dexmedetomidine 1 μg/kg with normal saline 5 ml.
  Other Names: Local anesthetic
  Arms: Bupivacaine + Dexmedetomidine group

SUMMARY:
For patients with symptomatic cholelithiasis, laparoscopic cholecystectomy (LC) is a customary procedure for treatment these days. After LC, patients may experience considerable pain. This study was performed with the objective of comparing the mean duration of analgesia of intraperitoneal bupivacaine with dexmedetomidine to intraperitoneal bupivacaine alone in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender
* Aged between 20 and 70 years
* ASA (American Society of Anesthesiologists Classification) physical status I and II
* Undergoing Laparoscopic Cholecystectomy under general anesthesia

Exclusion Criteria:

* Patients sensitive to local anesthetics
* Patients with acute cholecystitis, choledocholithiasis, or ascending cholangitis (temperature≥38.6°C, serum bilirubin≥1.2mg/dl, and ultrasound showing common bile duct diameter of ≥1cm).
* Patients with uncontrolled diabetes (FBS≥110 mg/dl)
* Uncontrolled blood pressure (SBP≥140 mmHg)
* Ischemic heart disease (EF≤40%)
* Pulmonary dysfunction (FEV≤70 percent of normal)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours
  The duration of postoperative analgesia was calculated as the time in minutes starting after the dressing of the patient in the operation room until the patient had a VAS≥3.

CONTACTS AND LOCATIONS:
Overall Officials: Qazi Anees, FCPS, Principal Investigator — Bahawal Victoria Hospital; Syed Shakeel Ahmed, FCPS, Principal Investigator — Shahida Islam Teaching Hospital
Locations (1):
- Quaid-e-Azam Medical College, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable request